CLINICAL TRIAL: NCT03900793
Title: A Phase I/Ib Study of Losartan in Combination With Sunitinib in the Treatment of Pediatric and Adult Patients With Relapsed or Refractory Osteosarcoma
Brief Title: Losartan + Sunitinib in Treatment of Osteosarcoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Cancer League of Colorado (Other); Colorado State University (Other); Swim Across America (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 18-2740.cc; NCI-2019-06119 (Other: CTRP)
Record Dates: First submitted 2019-03-12; First posted 2019-04-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Osteosarcoma
Keywords: Pediatrics; Adults; Phase 1; Losartan; Sunitinib; Maximum Tolerated Dose; Recommended Phase 2 Dose
MeSH Terms: conditions — Osteosarcoma | interventions — Losartan; Sunitinib

STUDY DESIGN:
Intervention Model Description: Dose escalation for Phase 1 with dose levels described in Arms and interventions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dose Escalation and Expansion (Experimental): Part 1: This is a study escalating doses (Dose level 1-3) of losartan on a continuous daily dosing schedule and sunitinib (escalating on dose level 4) on a daily dosing with 4 weeks on, 2 weeks off. A cycle of therapy is 6 weeks (42 days).Dosing will be performed based on body surface area (BSA). This portion of the study uses a 3+3 design (i.e. cohort sizes of 3 patients for the first and second cohort at each dose level).
  Part 2: Once the Maximally Tolerated Dose (MTD) has been determined, 12 patients will enroll to the expansion cohort. These patients will receive the MTD as long as less then 33% of patients experience dose-limiting toxicities.
  Interventions: Drug: Losartan; Drug: Sunitinib

INTERVENTIONS:
Drug: Losartan — Losartan will be administered orally daily on days 1-42 (6 weeks) with dose level assignments. Dosing will be performed based on weight in kilograms and rounded to the nearest 12.5 mg (half of 25 mg tablet). Dose level 1 dosing will not exceed 50 mg daily, dose level 2 dosing will not exceed 100 mg daily, and dose level 3 dosing will not exceed 150 mg total daily (75 mg twice daily). Doses should be taken at approximately the same time daily and patients should fast for at least 4 hours prior to dosing
Drug: Sunitinib — Sunitinib will be administered orally daily on days 1-28 (4 weeks), followed by 14-day rest period (2 weeks). Dosing will be performed based on body surface area (BSA) in mg/m2. Sunitinib is given as capsules or liquid formulation. Doses should be taken at approximately the same time daily.
  Other Names: Sunitinib Malate

SUMMARY:
This study is a Phase 1/1b clinical trial that aims to determine the Maximally Tolerated Dose of Losartan and Sunitinib Combination Therapy. Patients will first be accrued to the Dose Escalation phase of the study, using a 3+3 design. Medication dosages will increase until a maximally tolerated dose is found. Patients will then be accrued to the Dose Expansion phase of the trial, where efficacy of pre-determined dose will be preliminarily assessed.

ELIGIBILITY:
Inclusion Criteria:

* 1. Provision to sign and date the consent form (if individual is a minor, provision of a parent or legal guardian to sign and date the consent form and provision of individual to provide assent for study).

  2. Stated willingness to comply with all study procedures and be available for the duration of the study.

  3. Male or female aged ≥ 10 years old. 4. Histologically confirmed osteosarcoma (at either original diagnosis or relapse) that has either recurred or progressed after at least one prior systemic therapy and for which no curative therapy exists.
* Patients with surface or periosteal osteosarcoma are not eligible.
* Patients with active CNS metastasis are not eligible. Previously treated CNS metastases which occurred 3 months or more prior, without evidence of active recurrence, are acceptable.

  5. Disease status
* Dose Escalation (Part A): Patients must have measurable or evaluable disease.
* Cohort Expansion (Part B): Patients with measurable or evaluable disease and those with completely resected disease are eligible.

  6. Performance status:
* ECOG performance status (≥18 years old) ≤ 2 or Karnofsky performance score (<18 years old)≥ 50.

  7. Prior Therapy:
* Patients must have fully recovered from the acute toxic effects of all prior anti-cancer therapy and must meet the following minimum duration from prior anti-cancer directed therapy prior to enrollment. If after the required timeframe, the numerical eligibility criteria are met (e.g., blood count criteria) the patient is considered to have recovered adequately.

  1. Cytotoxic chemotherapy or other anti-cancer agents known to be myelosuppressive. At least 21 days after the last dose of cytotoxic or myelosuppressive chemotherapy (42 days if prior nitrosourea).
  2. Anti-cancer agents not known to be myelosuppressive (e.g., not associated with reduced platelet or ANC counts): ≥ 7 days after the last dose of agent.

  i. Antibodies: ≥ 21 days must have elapsed from infusion of last dose of antibody, and toxicity related to prior antibody therapy must be recovered to Grade ≤ 1.

ii. Corticosteroids: ≥ 14 days must have elapsed since last dose of corticosteroid.

iii. Hematopoietic growth factors: ≥ 14 days after the last dose of a long- acting growth factor (e.g., pegfilgrastim) or 7 days for short-acting growth factor.

iv. Interleukins, Interferons and Cytokines (other than hematopoietic growth factors): ≥ 21 days after the completion of interleukins, interferon or cytokines (other than Hematopoietic Growth Factors).

v. Stem cell Infusions: Autologous stem cell infusion, including boost infusion: ≥ 42 days.

vi. Cellular Therapy: ≥ 42 days after the completion of any type of cellular therapy (e.g., modified T cells, NK cells, dendritic cells, etc.) vii. XRT/External Beam Irradiation including protons: ≥ 14 days after local XRT; ≥ 150 days after TBI, craniospinal XRT or if radiation to ≥ 50% of the pelvis; ≥ 42 days if other substantial bone marrow radiation.

* NOTE: Patients with history of cardiac irradiation with mean cardiac dose > 15 Gy are not eligible (see exclusion criteria).

  8. Adequate bone marrow function, defined as:
* Peripheral absolute neutrophil count (ANC) ≥ 750/mm3
* Platelet count ≥ 75,000/mm3 (transfusion independent, defined as not receiving platelet transfusions for at least 7 days prior to enrollment).
* Hemoglobin ≥ 8 g/dL (with or without transfusion) 9. Adequate renal function, defined as:
* Creatinine clearance or radioisotope GFR > 70 mL/min/1.73 m2 OR a serum creatinine based on age/gender.

  10. Adequate hepatic function, defined as:
* Total bilirubin ≤ 1.5 x upper limit of normal (ULN) for age
* SGPT (ALT) ≤ 135 U/L. For the purpose of this study, the ULN for SGPT is 45 U/L.
* Serum albumin ≥ 2.8 g/dL 11. Patients with ≥ trace protein on urinalysis at screening will be allowed to enroll in the study at investigator discretion. A baseline urine protein creatinine ratio (UPC) should be obtained for patients with ≥ trace protein on urinalysis for consideration regarding Section 6.3.7 dose modification requirements.

  12. Adequate cardiac function, defined as:
* Current cardiac ejection fraction > 50% by biplane Simpson method on echocardiogram
* QTc ≤ 480 ms 13. Patients with preexisting hyper- or hypothyroidism must be on a stable dose of medication.

  14. Ability to take and retain oral medications. NOTE: Medication can be administered via nasogastric or gastrostomy tube.

Exclusion Criteria:

1. Patients who underwent major surgery within 14 days prior to start of treatment are not eligible.

   NOTE: Core biopsy or central line placement are considered minor and are allowed within any time limitations.
2. Patients with uncontrolled coagulopathy or bleeding disorder, or any active bleeding (i.e., gastrointestinal or pulmonary) deemed to be clinically significant by investigator are not eligible.
3. Patients with history of pulmonary embolism or significant thromboembolic event with the preceding 28 days. Patients with thromboembolic events > 28 days before enrollment who are stable on or completed an anticoagulation course are eligible.
4. Patients with history of cardiac irradiation with mean cardiac dose > 15 Gy are not eligible.
5. Patients with symptomatic cardiac disease (i.e. New York Heart Association or Modified Ross Heart Failure Classification for Children > class 2) are not eligible.
6. Patients with any history of cardiac dysfunction including prior abnormal echocardiogram (ejection fraction < 50%), severe or unstable angina, peripheral vascular disease, congenital prolonged QTc syndrome, clinically significant cardiac arrhythmias, stroke, or myocardial infarction are not eligible.
7. Pregnancy

   * Pregnant or breast-feeding women will not be entered on this study because there is not yet available information regarding human fetal or teratogenic toxicities. Pregnancy tests must be obtained in females who are post-menarchal.
   * Males or females of reproductive potential may not participate unless they have agreed to practice 1 highly effective and 1 additional effective (barrier) method of contraception at the same time during the entire study treatment period and through 3 months after the last dose of study drug, or agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the subject. Patients who themselves or their partners have undergone female or male sterilization do not require 2 methods of contraception. Highly effective methods are defined as those with <1% failure rate with perfect use and include: oral contraceptive pills (combined or progesterone only), intrauterine devices (IUD), hormonal implant or injection, contraceptive patch, and vaginal ring.
8. Concomitant medications:

   * Anti-hypertensives: Patients who cannot be controlled to goal blood pressure for gender/age are not eligible.
   * Corticosteroids: Patients receiving systemic corticosteroids are not eligible. > 14 days must have elapsed since last systemic corticosteroid. Note: patients using topical or inhaled corticosteroids are eligible.
   * Investigational Drugs: Patients currently receiving another investigational drug are not eligible.
   * Anti-cancer agents: Patients currently receiving other anti-cancer agents are not eligible.
   * Drug interactions: Patients who require treatment with medications that are strong inhibitors or inducers of CYP3A4 or inhibitors of CYP2A9 or have received these medications in the 7 days prior to enrollment, are not eligible. Patients who require treatment with enzyme inducing anticonvulsants are not eligible.
   * Medications that prolong QTc: Patients who require treatment with medications known to prolong QTc are not eligible

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 41 (Estimated)
Dates: Start 2019-08-26 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Assessment of Dose-Limiting Toxicities of Losartan and Sunitinib Combination | Beginning of study to end of study, up to 4 years
  Assessment of Dose-Limiting Toxicities (DLTs) according to the Common Terminology Criteria for Adverse Events (CTCAE) version 5 to assess the safety of the combination
Maximally Tolerated Dose of Losartan and Sunitinib | Beginning of study to end of study, up to 4 years
  The MTD will be defined as the dose level below that at which 1/3 or 2/6 patients experience DLTs.
Recommended Phase 2 Dose of Losartan and Sunitinib | Beginning of study to end of study, up to 4 years
  The dose than less that 33% of patients experience DLTs.

SECONDARY OUTCOMES:
Pharmacokinetics of Losartan and Sunitinib in Pediatric and Adult Patients: Maximum Peak Concentration | Days 1, 15, and 29 of Cycle 1 (Cycle length is 42 days)
  Determined through blood samples
Pharmacokinetics of Losartan and Sunitinib in Pediatric and Adult Patients: Time to Peak Concentration | Days 1, 15, and 29 of Cycle 1 (Cycle length is 42 days)
  Determined through blood samples
Pharmacodynamics of Losartan and Sunitinib in Pediatric and Adult Patients: CCL2-Mediated Chemotactic Index | Beginning of study to end of treatment, up to 2 years (up to 17 cycles and cycle length is 42 days)
  Determined through a monocyte mitigation assay and reported as a change in chemotactic index from baseline
Pharmacodynamics of Losartan and Sunitinib in Pediatric and Adult Patients: Plasma CCL2 Levels | Beginning of study to end of treatment, up to 2 years (up to 17 cycles and cycle length is 42 days)
  Assessed by Enzyme Linked Immunosorbent Assay (ELISA).
Pharmacodynamics of Losartan and Sunitinib in Pediatric and Adult Patients: CCR2+ Monocyte Population | Beginning of study to end of treatment, up to 2 years (up to 17 cycles and cycle length is 42 days)
  Assessed by Flow Cytometry
Preliminary Antitumor Activity of Losartan and Sunitinib in Pediatric and Adult Patients: Disease Control Rate (DCR) | Beginning of study, end of cycle 1 (each cycle is 6 weeks), and at the end of odd cycles (up to 17 cycles)
  Stable disease determined according to RECIST 1.1 criteria
Preliminary Antitumor Activity of Losartan and Sunitinib in Pediatric and Adult Patients: Disease Control Rate (DCR) | Beginning of study, end of cycle 1 (each cycle is 6 weeks), and at the end of odd cycles (up to 17 cycles)
  Partial response determined according to RECIST 1.1 criteria
Preliminary Antitumor Activity of Losartan and Sunitinib in Pediatric and Adult Patients: Disease Control Rate (DCR) | Beginning of study, end of cycle 1 (each cycle is 6 weeks), and at the end of odd cycles (up to 17 cycles)
  Complete response determined according to RECIST 1.1 criteria
Preliminary: Progression Free Survival (PFS) | Beginning of study, end of cycle 1 (each cycle is 6 weeks), and at the end of odd cycles (up to 17 cycles)
  Determined according to irRECIST criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Kelly Faulk, MD, Principal Investigator — Children's Hospital Colorado
Locations (4):
- United States (4):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Children's Hospital Colorado, Aurora, Colorado
  - University of Colorado Hospital, Aurora, Colorado
  - Children's Hospital of Atlanta, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: No